CLINICAL TRIAL: NCT04050748
Title: Comparison of Tendon Lengthening With Traditional vs. Accelerated Rehab Following Achilles Tendon Repair: A Prospective Randomized Controlled Trial
Brief Title: Achilles Tendon Lengthening With Traditional vs. Accelerated Rehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Toufic R. Jildeh, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 37283847
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Achilles Tendon Rupture

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Rehabiliation (Placebo Comparator): 6 weeks of non-weight bearing in addition to basic stretching exercises.
  Interventions: Procedure: Achilles tendon repair
- Accelerated Rehabilitation (Active Comparator): Patients will be non-weight bearing for 2 weeks. After 2 weeks patients were transitioned to a boot with two heel wedges and were weight bearing as tolerated. At 4 weeks, patients were transitioned to one wedge, and at 6 weeks patients were weight bearing as tolerated in a flat shoe. Each heel wedge was ¾ inch tall. After 6 weeks, patient's in both groups underwent identical rehab regimens per protocol
  Interventions: Procedure: Achilles tendon repair

INTERVENTIONS:
Procedure: Achilles tendon repair — Patients will be undergoing achilles tendon repair

SUMMARY:
The purpose of this study is to evaluate the surgically repaired tendon of a ruptured achilles tendon. We will investigate fixation slippage and tendon creep and correlate how these post-repair findings can contribute to outcomes of tendon repairs.

DETAILED DESCRIPTION:
pture of the Achilles tendon is a relatively common injury among athletes involved in sports which require rapid direction changes and accelerations, such as soccer, sprinting, and basketball. Approximately 80% of ruptures occur during recreational sports, but it can also occur in sedentary individuals. An increase in recreational sport involvement has coincided with an increase in Achilles tendon ruptures. The most common age group for this injury is between 30 and 40 years old, and it is more likely to occur in males. It is thought that rupture in this age group is highest due to the co-occurrence of competitive sports and age- related degenerative changes.

Tendons changes occur as we age. There is decreased collagen density and fewer cross links, which alters the integrity of the tendon and its sheath. These changes, in addition to repetitive microtrauma, can cause the Achilles tendon to become calcified and thickened. Alteration in the elasticity of the tendon can set the stage for a rupture during abrupt increases in training intensity or during competitions.

The Achilles tendon is the largest tendon in the body, and it receives its blood supply from the gastroc- soleus complex. The blood supply is weakest between 2cm and 6cm from the tendon's insertion on the calcaneus, which is also the region where it is most likely to rupture.

The current recommendation for acute Achilles rupture is surgical repair, but there is no consensus regarding surgical versus nonsurgical treatment (immobilization, rehab, etc.). Surgical repair is thought to reduce the rates of re-rupture but also cause an increased risk of complications. There does not appear to be a difference in pre-injury activity levels between the two methods.

Tendons have excellent healing potential when the torn ends are reasonably approximated. Optimal tendon healing depends on surgical apposition and mechanical stabilization of the tendon ends. Once a tendon has been repaired, the suture material holds the tendon ends together, allowing fibroblasts to produce sufficient amounts of collagen to form a tendon callus.

In contrast with approximated tears, neglected ruptures with retraction of the proximal portion of the tendon heal with scar tissue, resulting in a lengthened, weakened musculotendinous unit. Poor muscle function will result without restoration of normal tendon length. Studies of tendon healing have indicated that early controlled motion and tensile stress applied to a repaired tendon promote earlier organization and remodeling of collagen fibers, decreased scar tissue, and increased strength compared with tendon immobilization.

Previous studies involving Rotator cuff repairs and ACL ligament reconstructions have employed the use of Tantalum Beads and roentgen stereophotogrammetric analysis to evaluate the creep or stretch of repaired soft tissue. These studies show that there appears to be soft tissue stretch/creep that occurs as tendon and ligament repairs/reconstructions heal. A surgeon's knowledge of how a repaired soft tissue will deform or stretch will be an undoubted asset to patient care and management. This knowledge will be invaluable for the surgeon in regards to appropriately preparing a tendon for repair, directly repairing the tendon and appropriately tensioning of the repair. It will also give valuable information for rehabilitation protocols and activity limitations post-operatively.

The safety of tantalum material has well been described in the orthopaedic literature. It is currently used in implants ranging from cervical spinal fusions to femoral rods without side effects.

Recently a prospective study looking at creep in rupture biceps tendons has been completed our institution. This study will use stereophotogrammetric analysis to expand our investigations to include Achilles tendon.

ELIGIBILITY:
Inclusion Criteria:

- Patients with an acute tendon rupture less than 6 weeks were included in this study.

Exclusion Criteria:

- Underwent any additional concomitant procedures or tendon transfers, sustained prior ruptures, or had a chronic rupture.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Repair site lengthening | 2 years
  Intratendinous and repair site lengthening were determined

SECONDARY OUTCOMES:
Achilles Tendon Total Rupture Score | 2 years
  measure symptoms and physical activity levels after being treated for a complete Achilles tendon rupture

CONTACTS AND LOCATIONS:
Locations (1):
- Health Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Okoroha KR, Ussef N, Jildeh TR, Khalil LS, Hasan L, Bench C, Zeni F, Eller E, Moutzouros V. Comparison of Tendon Lengthening With Traditional Versus Accelerated Rehabilitation After Achilles Tendon Repair: A Prospective Randomized Controlled Trial. Am J Sports Med. 2020 Jun;48(7):1720-1726. doi: 10.1177/0363546520909389. Epub 2020 Mar 23. PMID 32203675